CLINICAL TRIAL: NCT00848367
Title: Optimizing Outcomes for Binge Eating, Depression and Weight Loss for Obese Women With Binge Eating Disorder by Matching to Group Psychological Treatments Based on Level of Attachment Anxiety
Brief Title: Binge Eating Disorder Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007254-01H
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High attachment anxiety condition (Experimental): 16 weeks of Group Psychodynamic Interpersonal Psychotherapy for patients with Binge Eating Disorder, matching them by attachment anxiety dimensions in order to enhance the impact of the therapy. It is hypothesized that by optimally matching patients to groups, they will have better clinical and health outcomes.
  Interventions: Behavioral: Group Psychodynamic Interpersonal Psychotherapy
- Low attachment anxiety condition (Experimental): 16 weeks of Group Psychodynamic Interpersonal Psychotherapy for patients with Binge Eating Disorder, matching them by attachment anxiety dimensions in order to enhance the impact of the therapy. It is hypothesized that by optimally matching patients to groups, they will have better clinical and health outcomes.
  Interventions: Behavioral: Group Psychodynamic Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Group Psychodynamic Interpersonal Psychotherapy — This intervention will consist of 16 weekly 90 minute sessions of Group Psychodynamic Interpersonal Psychotherapy (GPIP). GPIP was developed and empirically tested in a randomized controlled trial (RCT) at our Centre. GPIP will be preceded by an individual pre-group preparation session conducted by a psychologist trained in GPIP to orient the patient to the therapy. Patients are given a rationale for the treatment.

SUMMARY:
The main objective of the proposed study is to determine whether the effectiveness of a group therapy treatment for Binge Eating Disorder (BED) is improved and attrition reduced by optimally matching women with BED who have high attachment anxiety to Group Psychodynamic Interpersonal Psychotherapy (GPIP). This study represents the next phase in a program of research stemming from a previously conducted randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

•Overweight Women 18 years of age or older who binge eat at least twice per week for the past month.

Exclusion Criteria:

* unable speak English
* history of an eating disorder other than Binge Eating Disorder
* concurrent Diagnostic and Statistical Manual-IV (DSM-IV) diagnosis of bipolar disorder, psychosis, drug or alcohol problem
* pregnant or planning on becoming pregnant within the next year
* are currently or plan to become enrolled in a weight loss program within the next year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Tasca, Ph.D.C.Psych, Principal Investigator — University of Ottawa, Ottawa Hospital-General Campus
Locations (1):
- Regional Centre for the Treatment of Eating Disorders, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Tasca GA, Ritchie K, Demidenko N, Balfour L, Krysanski V, Weekes K, Barber A, Keating L, Bissada H. Matching women with binge eating disorder to group treatment based on attachment anxiety: outcomes and moderating effects. Psychother Res. 2013;23(3):301-14. doi: 10.1080/10503307.2012.717309. Epub 2012 Aug 24. PMID 22920044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were self-referred from advertisements distributed around Ottawa and surrounding area, or referred from the Regional Center for the Treatment of Eating Disorders at The Ottawa Hospital (Sept. 2007 to Mar.2009).
Groups:
- Low Attachment Anxiety Condition: In our study sample, the range of scores for the Need for Approval subscale of the Attachment Style Questionnaire was 1.86-5.71 (the possible range of this subscale is 1-7). Participants in this group scored lower than the cut off of 3.59 on the Need for Approval subscale of the Attachment Style questionnaire. They were assigned to therapy groups homogeneously composed of participants with low attachment anxiety (i.e. others that scored below the cut off). The type of therapy administered to this group was Group Psychodynamic Interpersonal Psychotherapy (GPIP; Tasca, G., Mikail, S. & Hewitt, P. Group Psychodynamic Interpersonal Psychotherapy: A Manual for Time Limited Treatment of Binge Eating Disorder. (2002).) Participants received 16 weekly 90 minute sessions of GPIP from a male or female therapist.
- High Attachment Anxiety Condition: In our study sample, the range of scores for the Need for Approval subscale of the Attachment Style Questionnaire was 1.86-5.71 (the possible range of this subscale is 1-7). Participants in this group scored greater than the cut off of 3.59 on the Need for Approval subscale of the Attachment Style questionnaire. They were assigned to therapy groups homogeneously composed of participants with high attachment anxiety (i.e. others that scored above the cut off). The type of therapy provided was called Group Psychodynamic Interpersonal Psychotherapy (GPIP; Tasca, G., Mikail, S. & Hewitt, P. Group Psychodynamic Interpersonal Psychotherapy: A Manual for Time Limited Treatment of Binge Eating Disorder. (2002).) Participants received 16 weekly 90 minute sessions of GPIP from a male or female therapist.
Period: Overall Study
Arm/Group | Low Attachment Anxiety Condition | High Attachment Anxiety Condition
Started | 52 | 50
Completed | 43 | 41
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- High Attachment Anxiety Condition: These participants scored greater than the cut off of 3.59 on the Need for Approval subscale of the Attachment Style questionnaire. They were assigned to therapy groups homogeneously composed of participants with high attachment anxiety.
- Low Attachment Anxiety Condition: These participants scored lower than the cut off of 3.59 on the Need for Approval subscale of the Attachment Style questionnaire. They were assigned to therapy groups homogeneously composed of participants with low attachment anxiety.
- Total: Total of all reporting groups
Arm/Group | High Attachment Anxiety Condition | Low Attachment Anxiety Condition | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 49 | 99
  >=65 years | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.29 (10.54) | 46.23 (12.67) | 44.32 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Binge Eating in the Past 28 Days
Time Frame: Pre and Post treatment, 6 months and 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Attachment Anxiety Condition | Low Attachment Anxiety Condition
Number analyzed (Participants) | 41 | 43
days
  Freq. of binge eating in the Past 28 days: Pre | 16.06 (6.57) | 14.48 (4.69)
  Freq. of binge eating in the Past 28 days: Post | 6.26 (6.45) | 7.40 (8.18)
  Freq. of binge eating in the Past 28 days: 6mo | 6.40 (8.66) | 6.56 (8.49)
  Freq. of binge eating in the Past 28 days: 12mo | 5.67 (6.14) | 4.10 (5.03)

2. Secondary Outcome: Depression Symptoms
Description: Early response to treatment is indicated by a reduction in depression symptoms measured by The Beck Depression Inventory II (BDI-II; Beck, Steer, & Brown, 1996). The BDI-II is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The range for this scale is 0-63. Higher scores represent more depressive symptoms. We included cases that were missing up to 8 missing items and calculated scores for participants with missing items by taking the weighted mean and multiplying by 21.
Time Frame: Pre and Post treatment, 6 months and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Attachment Anxiety Condition | Low Attachment Anxiety Condition
Number analyzed (Participants) | 50 | 52
units on a scale
  Depression Symptoms: Pre | 25.82 (10.58) | 16.42 (10.49)
  Depression Symptoms: Post | 15.51 (11.48) | 10.26 (8.31)
  Depression Symptoms: 6 month | 12.62 (9.52) | 8.30 (7.08)
  Depression Symptoms: 12 month | 17.32 (9.78) | 9.75 (10.26)

ADVERSE EVENTS:
Description: We have written 0 as the Total Number of Participants at Risk since the trial consists of group therapy to which there are no risks associated.
Arm/Group | High Attachment Anxiety Condition | Low Attachment Anxiety Condition
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No